CLINICAL TRIAL: NCT00502554
Title: Extracorporeal Photopheresis in Patients With Bronchiolitis Obliterans Syndrome (BOS) After Lung Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient patient recruitment and ECP capacity
Sponsor: Hannover Medical School (Other)
Collaborators: Therakos (Industry)
Responsible Party: Department for Respiratory Medicine, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4584
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2008-05

CONDITIONS: Bronchiolitis Obliterans
Keywords: lung function; FEV1
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Observation with standard care (macrolides, exercise, oxygen therapy etc.) alone.
  Interventions: Procedure: photopheresis
- 2 (Active Comparator): 2-day cycles of photopheresis every 3 weeks for 3 months
  Interventions: Procedure: photopheresis

INTERVENTIONS:
Procedure: photopheresis — 2-day cycles of photopheresis every 3 weeks for 3 months
  Other Names: photopheresis by Therakos

SUMMARY:
Investigation of photopheresis as new therapy regimen in patients with bronchiolitis obliterans syndrome after lung transplantation in a controlled, randomized study

DETAILED DESCRIPTION:
Bronchiolitis obliterans syndrome is the major cause of mortality after lung transplantation. 5 years after lung transplantation about 50% of all patients have this syndrome. There are nearly none therapy options. Besides effective therapy of any gastrooesophageal reflux and an oral medication with azithromycin none further regimens are known. Photopheresis could show in several studies a benefit for patients with gvhd after bone marrow transplantation or for chronic rejection after any other solid organ transplantation. Just little case reports could show beneficial effect in patients with bos after lung transplantation.

This is the first controlled, randomized study with patients with bos after lung transplantation to investigate the effectiveness of this therapy in that patients.

ELIGIBILITY:
Inclusion Criteria:

* Single/Double lung transplantation
* at least 6 months after lung transplantation
* bronchiolitis obliterans syndrome, Stadium > 1 (nach ISHLT 2001, FEV1 <80% Best), none other reason for worsening lung function (eg acute rejection, infection, extrapulmonary reasons, airway obstruction)
* none gastroesophageal reflux
* medication for > 3 months with Azithromycin with further decrease of FEV1, MEF 25-75
* bioptic prove that there is no acute rejection
* no improvement under steroid pulse therapy

Exclusion Criteria:

* tumor or hematologic disease
* acute rejection
* respiratory insufficiency (O2>2l/min, pCO2 >50 mm Hg)
* weight < 40 kg
* acute infection
* colonization with multiresistant pathogens

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
FEV1 stabilisation | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Fuehner Thomas, Doctor, Principal Investigator — Department Pneumology
Locations (2):
- Germany (2):
  - Department Pneumology, Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Dep. Pneumology, Hanover, Lower Saxony